CLINICAL TRIAL: NCT00898872
Title: Central Lymphoma Repository Tissue Procurement Protocol for Relapse or Recurrent Disease
Brief Title: SWOG-9245 Collecting and Storing Tissue Samples From Patients With Relapsed or Recurrent Non-Hodgkin Lymphoma After Treatment on a Southwest Oncology Group Clinical Trial
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000455162; SWOG-9245 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Lymphoma
Keywords: recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; Waldenström macroglobulinemia; adult nasal type extranodal NK/T-cell lymphoma; recurrent childhood grade III lymphomatoid granulomatosis; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; childhood Burkitt lymphoma; childhood nasal type extranodal NK/T-cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Extranodal NK-T-Cell; Dendritic Cell Sarcoma, Interdigitating | interventions — Cryopreservation

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: cryopreservation

SUMMARY:
RATIONALE: Collecting and storing samples of tissue from patients with non-Hodgkin lymphoma to study in the laboratory may help the study of cancer in the future.

PURPOSE: This laboratory study is collecting and storing tissue samples from patients with relapsed or recurrent non-Hodgkin lymphoma after treatment on a Southwest Oncology Group (SWOG) clinical trial.

DETAILED DESCRIPTION:
OBJECTIVES:

* Acquire fresh snap-frozen lymphoma tissue from patients with relapsed or recurrent non-Hodgkin lymphoma after treatment on a Southwest Oncology Group (SWOG) clinical trial.
* Establish a standard set of procedures for routine acquisition, banking, and study of lymphoma tissues within the SWOG.
* Use repository tissue to establish clinical correlations via presently activated phenotyping studies and future projected molecular studies assessing specimen DNA and RNA status.
* Examine the biology of therapy failure in relationship to changes in pretreatment and post-treatment immunophenotypic data.

OUTLINE: This is a multicenter study.

Tissues collected at biopsy are snap-frozen and archived for future molecular and genetic studies.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of relapsed or recurrent non-Hodgkin lymphoma (NHL)
* Previously registered on 1 of the following SWOG clinical trials for previously untreated NHL:

  * SWOG-8410
  * SWOG-8503
  * SWOG-8508
  * SWOG-8516
  * SWOG-8736
  * SWOG-8809
  * SWOG-8907
  * SWOG-8954
  * SWOG-9125
  * SWOG-9240
  * SWOG-9320
  * SWOG-9349
  * SWOG-9432
  * SWOG-9501
  * SWOG-9703
  * SWOG-S9704
  * SWOG-9800
* Tissue samples of relapsed or recurrent disease available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who consented to SWOG 9245 for banking
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 1993-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Acquisition of snap-frozen lymphoma tissues | July 2011

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Grogan, MD, Study Chair — University of Arizona; Thomas P. Miller, MD, Study Chair — University of Arizona; Richard I. Fisher, MD, Study Chair — James P. Wilmot Cancer Center
Locations (82):
- United States (82):
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Willamette Falls Hospital, Oregon City, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - McLeod Regional Medical Center, Florence, South Carolina
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming